CLINICAL TRIAL: NCT02210884
Title: Effects of Maternal Vitamin D Supplementation on Markers of Vitamin D Status and Related Infant and Maternal Outcomes in Southern Ethiopia
Brief Title: Maternal Vit D Supplements & Infant and Maternal Biomarkers & Outcomes in Southern Ethiopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oklahoma State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: HE1357
Record Dates: First submitted 2014-08-06; First posted 2014-08-07 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-02

CONDITIONS: Vitamin D Deficiency
Keywords: Vitamin D supplementation; Lactation; 25 hydroxyvitamin D; Breast feeding
MeSH Terms: conditions — Vitamin D Deficiency; Breast Feeding | interventions — Vitamin D; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D (Experimental): Weekly oral dose of 15,000 IU of Vitamin D3
  Interventions: Dietary Supplement: Vitamin D
- Placebo (Placebo Comparator): Placebo capsule containing no vitamin D
  Interventions: Dietary Supplement: Vitamin D

INTERVENTIONS:
Dietary Supplement: Vitamin D — Weekly oral supplementation with 15,000 IU vitamin D
  Other Names: Vitamin D3

SUMMARY:
Synthesis of vitamin D in the skin through the action of sunlight is a major source of vitamin D in parts of the world where foods are not fortified with the vitamin. Skin pigmentation (color), dress habits and season are some of the factors that limit sun exposure and affect vitamin D synthesis in the skin. Maternal vitamin D status is especially important to meet infant needs when newborns are not supplemented with vitamin D. In Ethiopia, vitamin D status of lactating women and infants and breast milk vitamin D concentration have never been assessed. The purpose of this study is to assess changes in maternal and infant markers of vitamin D status before and after vitamin D supplementation of the lactating mothers.

DETAILED DESCRIPTION:
Vitamin D is a vitamin that regulates calcium and phosphorous homeostasis and ensures proper mineralization of bone. Lactating women and infants are considered to be at risk of vitamin D deficiency due to increased needs for vitamin D and calcium. Stores of vitamin D acquired in utero and breast milk are the main sources of vitamin D for infants. Maternal vitamin D deficiency, exclusive breastfeeding, skin pigmentation and limited sun exposure are commonly seen in infants with rickets. However, the UV exposure, dress habits, traditional practices and other risk factors to vitamin D deficiency in Ethiopia have not been explored. This study aims to fill this research gap.

ELIGIBILITY:
Inclusion Criteria:

* Breastfeeding
* Available for enrollment within 2 weeks of delivery
* Residing in the study area in Ethiopia
* Apparently healthy

Exclusion Criteria:

* Self-reported chronic or acute disease condition
* Not breastfeeding
* Twin births

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Plasma 25(OH)D concentrations of lactating women | 3 months after enrollment
  Maternal plasma 25(OH) will be assessed at baseline and after three months of weekly supplementation with 15,000 IU vitamin D or placebo.
Plasma 25(OH)D concentrations of lactating women | 6 months after enrollment
  Maternal plasma 25(OH)D concentrations will be measured at 6 months after weekly supplementation with 15,000 IU vitamin D3 or placebo
Plasma 25(OH)D concentrations of lactating women | 1 year
  Maternal 25 (OH)D concentrations will be measured at 1 year after weekly supplementation with 15,000 IU of vitamin D or placebo
Plasma 25(OH) vitamin D of infants at 6 months of age | 6 months
  Plasma 25(OH) vitamin D of 6-month-old infants whose mothers received weekly doses of 15,000 IU vitamin D or placebo from time of enrollment
Plasma 25(OH) vitamin D of 1-year-old infants | 1 year
  Plasma 25(OH) vitamin D of 1-year-old infants whose mothers received weekly doses of 15,000 IU vitamin D or placebo from time of enrollment
Breast milk concentration of vitamin D | 3 months
  Breast milk concentration of vitamin D will be measured three months after enrollment in lactating women who have received 15,000 IU Vitamin D weekly or placebo.
Breast milk concentration of vitamin D | 6 months
  Breast milk concentration of vitamin D will be measured six months after enrollment in lactating women who have received 15,000 IU Vitamin D weekly or placebo.
Breast milk concentration of vitamin D | 1 year
  Breast milk concentration of vitamin D will be measured twelve months after enrollment in lactating women who have received 15,000 IU Vitamin D weekly or placebo.
Clinical Assessment of Infants for Rickets | 3 months
  Infants of mothers supplemented with 15,000 IU vitamin D weekly or with placebo will be clinically assessed for rickets
Clinical Assessment of Infants for Rickets | 6 months
  Infants of mothers supplemented with 15,000 IU vitamin D weekly or with placebo will be clinically assessed for rickets
Clinical Assessment of Infants for Rickets | 12 months
  Infants of mothers supplemented with 15,000 IU vitamin D weekly or with placebo will be clinically assessed for rickets

SECONDARY OUTCOMES:
Infant motor developmental milestones | Weekly for one year
  Progress toward standardized infant motor developmental milestones will be assessed weekly in infants whose mothers received 15,000 IU of vitamin D or placebo from time of study enrollment
Infant acute respirtory tract infections | Weekly for one year
  Incidence of infant acute respiratory tract infections will be assessed weekly in infants whose mothers received 15,000 IU of vitamin D or placebo from time of study enrollment
Infant anthropometry | Quarterly for one year
  Weight and length of infants will be assessed quarterly in infants whose mothers received 15,000 IU of vitamin D or placebo from time of study enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Barbara J Stoecker, PhD, Study Director — Oklahoma State University
Locations (1):
- Hawassa University, Awasa, Ethiopia

REFERENCES:
- [Derived] Girma M, Argaw A, Tilahun Tadesse B, Mulugeta B, Chowanadisai W, Stoecker BJ. Effects of weekly cholecalciferol supplementation of lactating mothers on vitamin D status, and infant growth and gross motor development: a randomized controlled trial in rural Ethiopia. Am J Clin Nutr. 2025 Nov;122(5):1306-1316. doi: 10.1016/j.ajcnut.2025.07.028. Epub 2025 Aug 5. PMID 40754215